CLINICAL TRIAL: NCT03148756
Title: Phase 2, Open-Label, Randomized, Multicenter Study to Compare the Efficacy and Safety of Dalbavancin to Standard of Care Antibiotic Therapy for the Completion of Treatment of Patients With Complicated Bacteremia or Documented Infective Endocarditis
Brief Title: Efficacy and Safety of Dalbavancin Compared to Standard of Care Antibiotic Therapy for the Completion of Treatment of Patients With Complicated Bacteremia or Infective Endocarditis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to business reasons.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAL-MD-09
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2018-09-10 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Endocarditis; Bacteremia
MeSH Terms: conditions — Endocarditis; Bacteremia | interventions — dalbavancin; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dalbavancin (Experimental): Dalbavancin 1500 mg, intravenous (IV) administration over 30 minutes on Day 1, and on Day 8.
  Interventions: Drug: Dalbavancin
- Standard of Care (Active Comparator): Antibiotic consistent with Standard of Care (SOC), based on baseline pathogen, for 4 to 6 weeks.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Dalbavancin — Dalbavancin 1500 mg, intravenous (IV) administration over 30 minutes on Day 1, and on Day 8.
  Arms: Dalbavancin
Drug: Standard of Care — Antibiotic consistent with Standard of Care (SOC), based on baseline pathogen, for 4 to 6 weeks.
  Arms: Standard of Care

SUMMARY:
This study will compare dalbavancin to standard of care (SOC) antibiotic therapy for the completion of therapy in patients with complicated bacteremia or infective endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of complicated bacteremia or infective endocarditis
* Gram-positive bacteremia at screening with methicillin-susceptible Staphylococcus aureus (MSSA), methicillin-resistant Staphylococcus aureus (MRSA) or Streptococci
* Treatment with standard of care antibiotics for 72 hours (h) - 10 days
* Defervescence for at least 24h and clearance of bacteremia from screening pathogen.

Exclusion Criteria:

* Embolic events
* History of prosthetic valve surgery, cardiac device or prosthetic joint
* Left-sided endocarditis due to Staphylococcus aureus (S. aureus)
* Large mobile vegetations (>10 mm) on mitral valves
* Perivalvular abscess
* Uncomplicated bacteremia due to S. aureus
* Gram-negative bacteria or fungi in blood cultures
* Heart failure associated with infective endocarditis [Left Ventricular Ejection Fraction (LVEF) <40%]
* Intravascular material or removable infection source not intended to be removed within 4 days postrandomization
* Planned valve replacement surgery within 3 days of randomization
* Refractory shock, significant hepatic insufficiency or severe leukopenia [Absolute Neutrophil Count (ANC) < 500 cells/mm^3]
* Known osteomyelitis
* Hypersensitivity to dalbavancin or other drugs in glycopeptide class
* Infection with enterococci, coagulase-negative staphylococci, or with organism not susceptible to dalbavancin or vancomycin
* Immunosuppression/immune deficiency
* Concomitant systemic antibacterial therapy for gram-positive infection other than that allowed in protocol
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Urania Rappo, MD, Study Director — Allergan
Locations (1):
- Midway Immunology and Research Center, Ft. Pierce, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalbavancin | Standard of Care
Started | 0 | 2
Completed | 0 | 1
Not Completed | 0 | 1
Not completed — Study Terminated | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalbavancin | Standard of Care | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at Day 84 in the Intent-to Treat (ITT) Population
Description: Clinical response was either success or failure. Success was defined as resolution of clinical signs and symptoms of complicated bacteremia or infective endocarditis (IE) such that no additional antibiotic therapy was required. Failure was defined as: ongoing signs and symptoms considered by the investigator to be related to complicated bacteremia or IE requiring additional antibacterial therapy or unplanned valve replacement, recurrent bacteremia, death during the study period up to Day 84 or discontinuation of the study medication due to an adverse event.
Time Frame: Day 84
Population: ITT Population included all randomized participants regardless of whether or not study treatment was received. No participants were enrolled in the Dalbavancin arm. Due to early termination of the study, 1 participant did not have clinical outcomes determined, but did have an early termination visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
Participants
  Success |  | 1
  Failure |  | 0

2. Secondary Outcome: Percentage of Participants With Clinical Outcome of Success at Day 42 in the ITT Population
Description: Clinical outcome was either success or failure. Success was defined as resolution of clinical signs and symptoms of complicated bacteremia or infective endocarditis (IE) such that no additional antibiotic therapy was required.
Time Frame: Day 42
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

3. Secondary Outcome: Percentage of Participants With Clinical Outcome of Success at Day 42 in the Clinically Evaluable (CE) Population
Description: as for outcome 2
Time Frame: Day 42
Population: CE Population included all participants in the mITT Population (all in the ITT who received ≥1 dose of study treatment) who met criteria for clinical evaluability. No participants were enrolled in the Dalbavancin arm. Due to early termination of the study, 1 participant did not have clinical outcomes determined, but did have a termination visit.
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

4. Secondary Outcome: Number of Participants With Day 84 Mortality in the Safety Population
Description: Day 84 mortality was measured by the number of deaths up to Day 84.
Time Frame: Day 84
Population: Safety Population included all randomized participants who received at least 1 dose of study treatment. No participants were enrolled in the Dalbavancin arm. Due to early termination of the study, 1 participant did not have clinical outcomes determined, but did have an early termination visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
Participants |  | 0

5. Secondary Outcome: Percentage of Participants With Clinical Outcome of Success at Day 84 in the CE Population
Description: Clinical outcome was either success or failure/relapse. Success was defined as resolution of clinical signs and symptoms of complicated bacteremia or infective endocarditis (IE) such that no additional antibiotic therapy was required.
Time Frame: Day 84
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

6. Secondary Outcome: Percentage of Participants With Clinical Outcome of Success by Pathogen at Day 42 in the ITT Population
Description: as for outcome 2
Time Frame: Day 42
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

7. Secondary Outcome: Percentage of Participants With Clinical Outcome of Success by Pathogen at Day 84 in the ITT Population
Description: as for outcome 2
Time Frame: Day 84
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

8. Secondary Outcome: Percentage of Participants With Clinical Outcome of Success by Pathogen at Day 42 in the CE Population
Description: as for outcome 2
Time Frame: Day 42
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

9. Secondary Outcome: Percentage of Participants With Clinical Outcome of Success by Pathogen at Day 84 in the CE Population
Description: as for outcome 2
Time Frame: Day 84
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

10. Secondary Outcome: Percentage of Participants With Microbiological Success by Pathogen at Day 42 in the ITT Population
Description: Microbiological outcome could be either microbiologic success or microbiologic failure. Microbiologic Success was defined as no further growth of baseline pathogen from blood cultures.
Time Frame: Day 42
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

11. Secondary Outcome: Percentage of Participants With Microbiological Success by Pathogen at Day 84 in the ITT Population
Description: as for outcome 10
Time Frame: Day 84
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

12. Secondary Outcome: Percentage of Participants With Microbiological Success by Pathogen at Day 42 in the CE Population
Description: as for outcome 10
Time Frame: Day 42
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

13. Secondary Outcome: Percentage of Participants With Microbiological Success by Pathogen at Day 84 in the CE Population
Description: as for outcome 10
Time Frame: Day 84
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

ADVERSE EVENTS:
Time Frame: Up to 84 Days
Description: There were no participants enrolled in the Dalbavancin arm. Due to the low number of participants enrolled at only 1 site, 0 participants are reported for SAEs due to the risk of identification of a person.
Arm/Group | Dalbavancin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalbavancin (N=0) | Standard of Care (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03148756/Prot_SAP_000.pdf